CLINICAL TRIAL: NCT06625008
Title: Impact of 3D-Printed Model on Shared Decision-Making and Anxiety in Patients Undergoing Surgery: the SEAD Pilot Randomized Trial
Brief Title: Preoperative 3D Models and Shared Decision-making
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Aimal Khan, Assistant Professor of Surgery, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 211314
Record Dates: First submitted 2024-09-18; First posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-09

CONDITIONS: Colorectal Cancer; Shared Decision Making; Anxiety; Informed Consent
Keywords: Colorectal cancer; 3D Model; Shared Decision Making; Preoperative anxiety; Patient knowledge; Informed Consent
MeSH Terms: conditions — Colorectal Neoplasms; Anxiety Disorders

STUDY DESIGN:
Masking Description: Masking was not performed as it was not feasible
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 3D-printed model arm (Experimental): Surgeons in this arm will use a 3D-printed modular human torso model with a magnetically detachable colon and rectum to teach patients about the anatomy and proximity of colonic segments undergoing surgery, potential surgical complications, and operative procedures during the pre-operative consent.
  Interventions: Other: 3D-printed model
- Standard care arm (No Intervention): Surgeons will employ the usual pre-operative counseling in this arm. This will include teaching patients about the anatomy, operative procedures, and potential surgical complications during the pre-operative consent using 2D images.

INTERVENTIONS:
Other: 3D-printed model — The Department of Radiology at Vanderbilt University Medical Center will create a 3D-printed human torso model that includes the colon, rectum, and a stoma on the abdominal wall. This model will be used to provide pre-operative counseling during the surgical consent for patients.
  Arms: 3D-printed model arm

SUMMARY:
The objectives of this study will be to quantify, using validated scales, the effects of 3D-printed models on shared decision-making and patient anxiety during the pre-operative consent and education process.

DETAILED DESCRIPTION:
In this single-center pilot cluster randomized controlled trial, the investigators will prospectively measure patient-reported outcomes on shared decision-making and change in anxiety and knowledge. This study will consist of two arms with at least 20 patients each. Six surgeons will be randomly assigned using the opaque sealed envelope method to counsel patients using a modular 3D-printed model or providing standard care during pre-operative clinic visits. The eligibility criteria for the control and investigational arms will be standardized. The biostatistician will use Student t-tests to compare mean scores and ANCOVA to compare the change in mean scores after the pre-operative clinic visit.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be >18 years
* Patients scheduled for surgical intervention that would involve partial or complete resection of the colon and/or rectum

Exclusion Criteria:

* Patients requiring complex surgical reconstruction of organs other than the colon and/or rectum

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Shared decision making | Within 30 minutes after the preoperative counselling session.
  Quantify and compare patient perception of involvement in decision-making in either arm, measured by the validated Shared Decision Making (SDM-Q9) tool.

SECONDARY OUTCOMES:
Change in patient anxiety | Within 30 minutes before and 30 minutes after the preoperative counselling session.
  Quantify and compare patient anxiety levels before and after the pre-operative consent, measured by the validated State-Trait Anxiety Inventory (STAI-6) among the study arms.
Change in patient knowledge using a self-developed questionnaire | Within 30 minutes before and 30 minutes after the preoperative counselling session.
  Using a self-developed questionnaire to quantify and compare patient knowledge of the essential aspects of anatomy, disease, and surgical procedure covered in preoperative counseling to understand how patient knowledge improves with counseling and compares between the study arms.

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khan A, Sellyn GE, Ali D, Moazzam Z, Samaras H, McChesney SL, Hopkins MB, Ford MM, Muldoon RL, Geiger TM, Martin D, Chu DI, VanKoevering KK, Hawkins AT. Three-Dimensional-Printed Models and Shared Decision-Making: A Cluster Randomized Clinical Trial. JAMA Netw Open. 2025 Jun 2;8(6):e2513187. doi: 10.1001/jamanetworkopen.2025.13187. PMID 40459895